CLINICAL TRIAL: NCT00005703
Title: Hemostasis in Sickle Cell Disease--Infancy to Adulthood
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4310; R01HL055185 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-03

CONDITIONS: Anemia, Sickle Cell; Blood Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Hematologic Diseases

SUMMARY:
To assess in older children and adults with sickle cell disease (SCD) whether intrinsic activation (relevant to the origin of pain and acute inflammation) occurs only during vasocclusive crisis (VOC).

DETAILED DESCRIPTION:
BACKGROUND:

Investigations into hemostatic abnormalities associated with sickle cell disease have been numerous. The data suggested that thrombin generation and fibrin formation were increased during steady state, with conflicting data whether further activation occurred in vaso-occlusive crisis. Platelet activation during VOC occurred, with variable findings during steady state. A selective, concomitant evaluation of the hemostatic pathways i.e. intrinsic, tissue factor (TF) or extrinsic activation, fibrinolysis, and platelet-endothelial activation had not been reported. Neither had a longitudinal evaluation been performed in infants during the unique transition period when HbF levels fall from 70 to 80 percent to less than 10 percent.

The study was part of an initiative on "Coagulation, Platelets and Thrombosis in Sickle Disease Pathophysiology". The Request for Applications was released in October 1994.

DESIGN NARRATIVE:

The studies used appropriate 'negative' and 'positive' control groups. Studies included intrinsic markers [kininogen profiling, high molecular weight kininogen (HK) and low molecular weight kininogen (LK) cleavages, western blotting of HK and LK, and kallikrein-alpha2 macroglobulin; extrinsic markers [TF and factor V11a]; other activation and fibrinolytic markers [prothrombin F1.2, FPA, TAT, tPA, PAI-I, D-dimer and plasma alpha2 antiplasmin]; platelet- endothelial markers [evaluation of activation dependent epitopes]. Unequivocal demonstration of contact pathway activation during VOC provided a crucial link between VOC and its accompanying phenomenon including pain, and inflammation. Finally, the studies provided a unique perspective on the continuum of hemostatic changes that unfolded during the course of SCD, and those that developed as vascular insufficiencies supervened in the adult.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-07; Study Completion 1998-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Stuart — Thomas Jefferson University